CLINICAL TRIAL: NCT02975999
Title: Use of Vasopressin Following the Fontan Operation: Both Pilot and Multicenter Studies
Brief Title: Use of Vasopressin Following the Fontan Operation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRP-530
Record Dates: First submitted 2016-09-22; First posted 2016-11-29 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Pleural Effusion; Single-ventricle
MeSH Terms: conditions — Pleural Effusion; Univentricular Heart | interventions — Vasopressins; Arginine Vasopressin; Arginine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vasopressin (Experimental): Vasopressin at 0.4mU/kg/min
  Interventions: Drug: Vasopressin
- Normal saline (Placebo Comparator): Normal saline will be provided on a drip infusion to the selected group once coming off cardiopulmonary bypass following the Fontan operation.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Vasopressin — Vasopressin at dose of 0.4mU/kg/min will be started on the assigned group once coming off cardiopulmonary bypass following the Fontan operation.
  Other Names: Vasostrict, arginine
  Arms: Vasopressin
Drug: Normal Saline — Normal saline at starting dose of 0.4mU/kg/min will be started on the assigned group once coming off cardiopulmonary bypass following the Fontan operation.
  Other Names: Placebo
  Arms: Normal saline

SUMMARY:
The purpose of this pilot study is to prepare for a larger study to determine whether Vasopressin following the Fontan operation will decrease chest tube output and duration.

DETAILED DESCRIPTION:
A pilot randomized, double blinded clinical trial to evaluate the use of vasopressin following the Fontan operation.

Phase one of the study will be a single center pilot study and will be conducted at Advocate Children's Hospital, Oak Lawn IL. This will be a randomized and double blinded. Ten patients will be enrolled with five patients as control group and five receiving Vasopressin. Vasopressin levels will be obtained just prior to initiation of Vasopressin and 48 hours later in the pilot study. Safety and effect size will be evaluated after this pilot study.

Drug administration protocol:

Vasopressin at a dose of 0.4 mU/kg/min will be started on subjects in the study group while coming off cardiopulmonary bypass. The dose of Vasopressin will not be titrated. Study drug drip will infuse for 48 hours after which will be discontinued.

The placebo group will be receiving normal saline at the same rate of the vasopressin group. The treating physician will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 1.5-7 years old undergoing Fontan operation.

Exclusion Criteria:

* Patients with a planned fenestrated Fontan.
* Patients undergoing revision surgery for failing Fontan.
* Evidence of renal insufficiency prior to surgery defined by creatinine >1 mg/dl.
* Planned arch reconstruction at the time of the Fontan procedure

Ages: 18 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Penk, MD, Principal Investigator — Advocate Health
Locations (1):
- Advocate Children's Hospital, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vasopressin | Normal Saline
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vasopressin | Normal Saline | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 12
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6 (1) | 5 (1) | 5 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 2 | 6 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Chest Tube Drainage
Description: chest tube drainage until the day the chest tube is removed
Time Frame: From post operative day 0 through study completion, an average of 1 month
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Vasopressin | Normal Saline
Number analyzed (Participants) | 6 | 6
ml/kg | 686.83 (307.03) | 535.50 (140.29)

2. Secondary Outcome: Length of Hospital Stay
Description: Duration the patient remains in the hospital in days until the day of discharge home
Time Frame: From the day of the surgery (post operative day 0) through study completion, an average of 1 month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Vasopressin | Normal Saline
Number analyzed (Participants) | 6 | 6
days | 5 (1.7) | 4.5 (0.8)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 years.
Arm/Group | Vasopressin | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT02975999/Prot_SAP_000.pdf